CLINICAL TRIAL: NCT01246375
Title: Prevalence of Osteoporosis in Patients Who Uses Inhaled Steroids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Yehuda Schwartz, Tel Aviv medical center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-10-SY-454-CTIL
Record Dates: First submitted 2010-11-21; First posted 2010-11-23 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Dual energy X-ray absorptiometry — Device which measures bone density

SUMMARY:
The purpose of this research is to determine whether the prevalence of osteoporosis is greater in patients who suffer from Chronic obstructive pulmonary disease (COPD) or Asthma disease and uses inhaled steroids.

ELIGIBILITY:
Inclusion Criteria:

1. Man at the minimum age of 60 years.
2. Diagnosed with Chronic Obstructive Pulmonary disease (COPD) or Asthma disease.
3. Usage of the following corticosteroids at the minimal doses indicated, for at least 3 years:

Seretide 250/50 mcg Symbicort 320/9 mcg 5.No Diagnosis of thyroid irregularity 6.No diagnosis/treatment for Osteoporosis.

Exclusion Criteria:

1. Usage of systemic steroids more than once during the 12 months prior to the study.
2. Usage of systemic steroids during the month prior to the study.
3. Usage of inhaled steroids in order to treat any other disease except Chronic Obstructive Pulmonary Disease (COPD) or Asthma.

Ages: 60 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Osteoporosis | 3 month
Diagnosis of Osteoporosis | 3

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Schwartz, M.D, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv medical center, Tel Aviv, Israel, Israel